CLINICAL TRIAL: NCT02633657
Title: A Multicenter, Open-label, Single-dose Pharmacokinetic and Safety Evaluation of HORIZANT (Gabapentin Enacarbil Extended-release Tablets) in Adolescents Aged 13 to 17 Years Old With Moderate-to-severe Primary Restless Legs Syndrome
Brief Title: A PK and Safety Evaluation of HORIZANT (Gabapentin Enacarbil) in Adolescents With Moderate-to-Severe Primary RLS
Acronym: RLS
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XP108
Record Dates: First submitted 2015-12-10; First posted 2015-12-17 (Estimated); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: RLS
Keywords: Restless Legs Syndrome; RLS
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Gabapentin; 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HORIZANT 300 mg (Experimental): HORIZANT 300 mg once daily
  Interventions: Drug: HORIZANT 300 mg

INTERVENTIONS:
Drug: HORIZANT 300 mg — HORIZANT 300 mg once daily
  Other Names: gabapentin enacarbil

SUMMARY:
The primary objective is to assess the pharmacokinetics (PK) of gabapentin following the single-dose administration of HORIZANT (Gabapentin Enacarbil) in adolescents (13 to 17 years of age) diagnosed with moderate-to-severe Primary Restless Legs Syndrome (RLS).

DETAILED DESCRIPTION:
One-treatment, 1-period study in adolescents (13 to 17 years of age) diagnosed with moderate-to-severe primary RLS. Patients will check-in at the clinical site in the evening of Day -1 or the morning of Day 0, and baseline safety assessments will be performed. On Day 0, after the review of these safety assessments and confirmation of eligibility, patients will receive a single oral 300 mg dose of HORIZANT with a meal (at approximately 6 AM). Study assessments will continue until approximately 14 hours (h) post dose, at which time patients will be discharged. Prior to discharge, patients will be advised not to drive a car or operate other complex machinery for at least 30 h after dosing; therefore, patients can remain at the clinical site overnight or can be escorted home. Patients will return to the clinical site for a follow-up visit 7 days (± 1 day) post dose.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adolescent patients, aged 13 to 17 years, diagnosed with RLS based on the IRLSSG consensus criteria, which is presented in Appendix 2.
2. Total RLS severity score of 15 or greater on the IRLS rating scale at screening.
3. Body weight greater than 33.4 kg and a healthy weight using age-based body mass index (BMI) range 5th to 85th percentile. Appendix 3 contains BMI-for-age charts that can be consulted.
4. Negative pregnancy test for females of childbearing potential. Female patients of childbearing potential must agree to use one of the following acceptable birth control methods:

   1. intrauterine device in place for at least 3 months prior to dosing
   2. barrier methods (male condom, female condom, diaphragm or cervical cap) with spermicide for at least 30 days prior to dosing and throughout the study
   3. stable hormonal contraceptive (including oral, injection, or implants) for at least 3 months prior to dosing and throughout the study Female patients who normally abstain from sexual activity may be recruited providing they remain abstinent during the study, or if they become sexually active, they must agree to use effective methods of birth control as described above.
5. Male patients able to father a child must agree to use a barrier method (male condom, female condom, diaphragm or cervical cap) with spermicide for at least 30 days prior to dosing and throughout the study. Male patients who normally abstain from sexual activity may be recruited providing they remain abstinent during the study, or if they become sexually active, they must agree to use a barrier method as described above.
6. Signed patient/parent Institutional Review Board (IRB)-approved informed consent/assent form (as applicable) prior to any study procedures.

Exclusion Criteria:

1. History of allergy, hypersensitivity or intolerance to HORIZANT or any other gabapentin compounds.
2. Suffering from a movement disorder that could mimic or confound the accurate diagnosis of RLS (eg, Tourette's syndrome, tic disorder, periodic limb movement disorder [PLMD], sleep disorders).
3. Currently meet Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5) criteria for substance use disorder, or history thereof, within 12 months prior to dosing.
4. Current or past history of any significant psychiatric disorder including but not limited to depression (treatment with antidepressants), bipolar disorder or schizophrenia.
5. History of suicidal behavior or suicidal ideation as indicated by the Columbia Suicide Severity Rating Scale (C-SSRS), administered at screening (the questionnaire is presented in Appendix 4), and as per investigator's judgment.
6. History of seizure disorder or at increased risk for development of a seizure disorder, including but not limited to complicated febrile seizure and history of significant head injury.
7. Medical condition or disorder that would interfere with the action, absorption, distribution, metabolism, or excretion of gabapentin enacarbil, or, in the investigator's judgment is considered to be clinically significant and may pose a safety concern, or, could interfere with the accurate assessment of safety or efficacy, or could potentially affect a patient's safety or study outcome.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2017-07-19 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from the time of dosing to the last measurable concentration (AUC0-tlast). | 0-14 hours
  AUCtlast
Area under the concentration-time curve from the time of dosing extrapolated to infinity (AUCinf) | 0-14 hours
  AUCinf
Percentage of AUCinf that is extrapolated from time of last measurable concentration to infinity (AUCextr%) | 0-14 hours
  % AUCinf
Maximum observed plasma drug concentration (Cmax) | 0-14 hours
  Cmax
Time to maximum concentration (Tmax) | 0-14 hours
  Tmax
Apparent elimination half-life (T1/2) | 0-14 hours
  T1/2
Apparent oral clearance (CL/F) | 0-14 hours
  CL/F
Apparent oral volume of distribution (Vd/F) | 0-14 hours
  Vd/F

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) | 7 days
  Columbia-Suicide Severity Rating Scale (C-SSRS)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Caras, MD, Study Director — Xenoport/Arbor Pharmaceuticals, LLC
Locations (4):
- United States (4):
  - Stanford Sleep Medicine Center, Redwood City, California
  - Pacific Research Network, St Louis, Missouri
  - SleepMed of South Carolina; SleepMed, Inc., Columbia, South Carolina
  - Vanderbilt University School of Medicine, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No